CLINICAL TRIAL: NCT06889571
Title: A Single-arm Feasibility Study of Nurse-supported Mobile App for Self-help CBT-I in Cancer Caregivers
Brief Title: Feasibility of a Nurse-Supported Mobile App for Self-Help CBT-I in Cancer Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yangxi Huang, Principal Investigator, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nurse-supported CBT-I 2025
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Cancer Caregivers
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nurse-Supported Mobile App for Self-Help CBT-I in Cancer Caregivers (Experimental)
  Interventions: Behavioral: Nurse-Supported Mobile App for Self-Help CBT-I

INTERVENTIONS:
Behavioral: Nurse-Supported Mobile App for Self-Help CBT-I — The intervention consists of two components: 1) a mobile app delivered 6-week self-help CBT-I program; and 2) Weekly nurse support session.

SUMMARY:
Study Goal The goal of this clinical trial is to evaluate whether a nurse-supported mobile app for self-help cognitive behavioral therapy for insomnia (CBT-I) is feasible for cancer caregivers and whether it can improve their sleep-related outcomes and overall well-being.

Main Questions

1. Feasibility:

   Can the intervention be successfully implemented in terms of recruitment, retention, adherence to the intervention protocol, safety, and participant satisfaction?
2. Preliminary Effects:

Does the intervention improve subjective sleep outcomes (e.g., insomnia severity, sleep quality, total sleep time, time in bed, sleep efficiency, wake after sleep onset, and sleep onset latency) as well as depressive symptoms, anxiety symptoms, fatigue, caregiver burden, and health-related quality of life?

What Participants Will Do i) Use a 6-week self-help CBT-I program delivered via a WeChat mini program. ii) Receive weekly nurse support sessions (up to 20 minutes each) for six weeks.

* These sessions may be conducted via phone calls or instant messaging, based on participant preference.
* Each session includes reviewing weekly progress, addressing any barriers to adherence, and planning next steps.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informal caregiver (e.g., family members, friends, or neighbors) who co-resides with and provides unpaid care for cancer survivors of any site or stage, with daily contact of at least 4 hours. If two or more caregivers are available for a cancer survivor, the one providing most of the daily care will be included.
* Able to understand the research procedures, and read and communicate in Chinese
* Able to use WeChat
* Insomnia severity index scores > 7

Exclusion Criteria:

* Another sleep disorder (e.g., obstructive sleep apnea, restless leg syndrome, rapid eye movement behavior disorder), besides insomnia, that is not adequately treated
* Psychotic disorders (e.g., bipolar disorder, schizophrenia); Suicidal ideation with intent and plan OR attempted suicide within the past 2 months
* Currently taking any psychotropic drugs (e.g., antidepressants, anxiolytics, sleep medications)
* Unstable or acute medical condition or condition requiring surgery in the next 6 months; Pregnancy; or Epilepsy
* Currently participating in any other interventional program
* Prior experience with CBT-I
* Night, evening, early morning or rotating shift work
* Currently caring for a cancer patient receiving hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Every month, up to 1 year
  The recruitment rate will be evaluated by the percentage of the target number of participants successfully recruited per month.
Retention rate | Post-intervention (i.e., at the end of the 6-week intervention period)
  The retention rate will be assessed by the percentage of recruited participants providing outcome data at post-intervention time point.
Adherence rate | Post-intervention (i.e., at the end of the 6-week intervention period)
  The adherence rate will be measured by the percentage of recruited participants who adhere to the proposed intervention, including reviewing sessions on the WeChat mini program and engaging in weekly nurse support sessions.
Participants' perspectives of acceptability and satisfaction | Post-intervention (i.e., at the end of the 6-week intervention period)
  The participants' perspectives of acceptability and satisfaction will be evaluated using eight adapted items from the Acceptability E-scale. Each item is rated on a 5-point Likert scale, with scores ranging from 1 to 5. The total score ranges from 8 to 40, with higher scores indicating greater acceptability and satisfaction with the intervention.
Adverse events | Throughout the study period (from baseline to post-intervention [i.e., at the end of the 6-week intervention period])
  All adverse events reported by the participants will be documented.
Participants' perceived experiences of the proposed intervention | Post-intervention (i.e., at the end of the 6-week intervention period)
  Participants' perceived experiences of the proposed intervention (e.g., intervention delivery, adherence, safety, and satisfaction) will be assessed through post-intervention qualitative interviews to provide a further understanding of the intervention's feasibility.

SECONDARY OUTCOMES:
Insomnia severity | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period）
  Insomnia severity will be assessed by Insomnia Severity Index (ISI). The ISI is a well-validated, 7-item scale designed to assess the severity of insomnia retrospectively over the past 2 weeks. Total scores range from 0 to 28, with higher scores indicating more severe insomnia symptoms.
Sleep patterns | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period)
  Sleep patterns (i.e., total sleep time [TST], time in bed [TIB], sleep efficiency [SE], wake after sleep onset [WASO], and sleep onset latency [SOL]) will be assessed using the Consensus Sleep Diary (CSD). The CSD is widely used to assess subjective sleep and help capture more subtle variations in sleep.
Sleep quality | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period)
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a widely used, 19-item questionnaire designed to measure various aspects of sleep quality over the past month. Scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Caregiver burden | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period)
  The caregiver burden will be evaluated by Zarit Burden Interview-12 (ZBI-12). The ZBI-12 is a widely used, 12-item shortened version of the original ZBI, designed to assess the subjective burden experienced by informal caregivers. Total scores range from 0 to 48, with higher scores indicating a greater level of caregiver burden.
Depressive symptoms | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period)
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a widely used, 9-item questionnaire designed to screen for, diagnose, monitor, and measure the severity of depression. Each item evaluates the frequency of depressive symptoms experienced over the past two weeks. Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.
Anxiety symptoms | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period)
  Anxiety symptoms will be assessed using the Generalized Anxiety Disorder-7 (GAD-7). This self-administered, 7-item questionnaire was designed as a screening tool and a severity measure for GAD. Each item asks about the frequency of anxiety symptoms over the past two weeks. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Fatigue | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period)
  Fatigue will be assessed using the Multi-Dimensional Fatigue Inventory (MFI). The MFI is a 20-item self-report questionnaire designed to measure five dimensions of fatigue (i.e., general fatigue, mental fatigue, physical fatigue, reduced activity, and reduced motivation). Total scores range from 20 to 100, with higher scores indicating greater levels of fatigue.
Health-related quality of life | T0 (Baseline): prior to the start of the intervention, T1 (6 weeks): Post-intervention (i.e., at the end of the 6-week intervention period)
  Health-related quality of life will be assessed using the five-dimension five-level European Quality of Life scale (EQ-5D-5L). The EQ-5D-5L is a standardized questionnaire designed to evaluate five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L score ranges from -0.39 to 1, with higher scores indicating better quality of life. Additionally, the EQ-5D-5L includes a Visual Analog Scale (VAS) for overall self-rated health status, with scores ranging from 0 to 100, where higher scores represent better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided